CLINICAL TRIAL: NCT02420483
Title: Lung Ventilation During Cardiopulmonary Resuscitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, DEMOSTHENES MAKRIS, ASS PROFESSOR CRITICAL CARE MEDICINE, University of Thessaly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49304 11/11/13
Record Dates: First submitted 2015-03-27; First posted 2015-04-17 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Ventilation During Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Cardiopulmonary resuscitation with measurement of tidal volume, airway pressure and flow by a pneumotachograph and airway, oesophageal pressure sensors
  Interventions: Other: Cardiopulmonary resuscitation chest compressions

INTERVENTIONS:
Other: Cardiopulmonary resuscitation chest compressions

SUMMARY:
The authors to measure passive tidal volumes generated during external chest compressions in order to determine whether chest compressions alone without any mechanical ventilatory support in cardiopulmonary resuscitation can provide adequate ventilation. The authors will study 25 volunteers who meet the following inclusion criteria: age 18-55 years, ASA I-II, candidates for surgical operation, who will receive general anesthesia. Patients who will be operated in the chest, who present musculoskeletal diseases, cardiopulmonary or vascular acute or chronic diseases, who had history of pneumothorax, of thromboembolism, osteoporosis, menopause, history of current rib or sternal or clavicle fractures, will be excluded. All eligible patients will enter the study and will receive general anesthesia and intubation according to treating doctors' decision.

Patients will be ventilated mechanically for 5 minutes to establish stable conditions. A pneumotachograph will be then connected to the ventilatory circuit so that respiratory efforts (volume, airway pressure and flow) can be continuously monitored at real time.

An esophageal catheter will be then inserted to monitor esophageal pressures and to provide data for lung mechanics calculation. Following the above procedures and before any surgical procedure, chest compressions will be performed to the patient by a senior anesthesiologist according to ERC guidelines of 2010 for 30 seconds.

Following chest compressions, patients will be evaluated for possible complications and after the establishment of stable conditions surgical procedures will follow. After the end of the surgical operation clinical and chest ultrasound evaluation will be performed.

Written inform consent will be obtained by all patients before procedures.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55 years
* ASA I-II
* candidates for surgical operation who will receive general anesthesia

Exclusion Criteria:

* surgical operation in the chest
* musculoskeletal diseases
* cardiopulmonary or vascular acute or chronic diseases
* history of pneumothorax
* thromboembolism
* osteoporosis menopause history of current rib or sternal or clavicle fractures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Tidal volume during cardiopulmonary resuscitation | 30 seconds
  Tidal volume will be assessed by a pneumotachograph (Hans Rudolf USA)

SECONDARY OUTCOMES:
Esophageal pressures during cardiopulmonary resuscitation | 30 seconds
  esophageal pressures will be assessed with an esophageal balloon-catheter that will be introduced via the nares while the patients is still awake and will be positioned at 40 cm from the nares. Correct positioning will be confirmed by the demonstration of negative pressure swings against an occluded airway.
Lung compliance before and at the end of cardiopulmonary resuscitation | 30 seconds
  Lung compliance will be assessed as the ratio of tidal volume change over transpulmonary pressure changes (subtracting oesophageal pressures from airway pressures) during tidal breathing (average of 10 breaths); oesophageal will be used as a measure of pleural pressures.

CONTACTS AND LOCATIONS:
Locations (1):
- Uh Larissa, Larissa, Thessaly, Greece